CLINICAL TRIAL: NCT07118839
Title: MDMA-Assisted Therapy for Veterans With PTSD and Alcohol Use Disorder: A Randomized Controlled Trial
Brief Title: MDMA-Assisted Therapy for Veterans With PTSD and Alcohol Use Disorder
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5603-R
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Post Traumatic Stress Disorder; Alcohol Use Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Alcoholism

STUDY DESIGN:
Intervention Model Description: This is a randomized study. Participants will be 1:1 randomized to receive either MDMA-AT or identical psychotherapy with active placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Full dose MDMA-Assisted Therapy (Experimental): Initial dose of 80 mg MDMA HCl administered orally at the start of each of three dosing sessions, possibly followed by a supplemental dose of 40 mg MDMA HCl 1.5 to 2 hours later. At dosing sessions 2 and 3, participants will be offered the option of taking a higher dose, 120 mg MDMA HCl, possibly followed by a supplemental dose of 60 mg MDMA HCl 1.5 to 2 hours later.
  Interventions: Drug: Full Dose MDMA; Behavioral: MDMA-AT
- Active Placebo dose MDMA-Assisted Therapy (Active Comparator): During the three Experimental Sessions, participants will receive the active placebo dose (one capsule) consisting of 40 mg MDMA HCl plus a second capsule containing an inactive placebo (indistinguishable weight placebo comprised entirely of mannitol and magnesium stearate), followed 1.5-2 hours later by the inactive placebo. The number of capsules comprising the initial dose (two) is consistent across both conditions.
  Interventions: Behavioral: MDMA-AT; Drug: Active Placebo Dose MDMA

INTERVENTIONS:
Drug: Full Dose MDMA — 3 MDMA dosing (Experimental) sessions: Session 1 - 80mg to 120mg MDMA HCl; Session 2 - 80mg to 180mg MDMA HCl; Session 3 - 80mg to 180mg MDMA HCl
  Arms: Full dose MDMA-Assisted Therapy
Behavioral: MDMA-AT — inner-directive psychotherapy will be conducted throughout the study; Lykos Therapeutics MDMA-AT Manual
Drug: Active Placebo Dose MDMA — 3 MDMA dosing (Experimental) sessions in which participants will receive 40mg MDMA HCl max at each session.
  Arms: Active Placebo dose MDMA-Assisted Therapy

SUMMARY:
The study investigators are conducting the first randomized placebo-controlled trial of MDMA-assisted therapy (MDMA-AT) with a comorbid sample of military Veterans with a co-occurring diagnosis of Alcohol Use Disorder (AUD) and Post-Traumatic Stress Disorder (PTSD). This novel experimental treatment package consists of three once-monthly Experimental Sessions of therapy combined with a divided-dose of MDMA HCl, along with non-drug preparatory and integrative therapy. The primary objective of the proposed project is to evaluate safety and clinical outcomes of MDMA-AT compared to identical psychotherapy with low dose ("active placebo") MDMA for the treatment of PTSD-AUD in military Veterans. The Primary Outcome measures, the Clinician Administered PTSD Scale (CAPS-5) and Inventory of Psychosocial Functioning (IPF), will evaluate changes in PTSD symptoms and psychosocial outcomes over time. Changes in drinking outcomes will also be evaluated (via the Timeline Followback, TLFB).

DETAILED DESCRIPTION:
The study will use a longitudinal design to conduct a randomized controlled trial of MDMA-AT for Veterans with PTSD-AUD. Eligible participants will complete an in-person baseline assessment, engage in MDMA-AT or identical psychotherapy with low dose ("active placebo") MDMA with clinicians trained by Lykos Therapeutics, and complete assessments at post-treatment, 3-, and 6-month follow-ups. For complete description of the investigational plan, please the attached Clinical Protocol.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study if all the following criteria apply:

Age

1. Are at least 18 years old at the time of signing the informed consent. Type of Participant and Disease Characteristics
2. Are currently enrolled in VA care.
3. Veterans must have initiated and discontinued (or completed) at least one first-line evidence-based treatment (EBT) for PTSD alone, for PTSD and AUD together, or for a dual-diagnosis condition, as documented in CPRS.
4. Are fluent in speaking and reading English.
5. At Baseline, meet past-year criteria for Alcohol Use Disorder as measured by the SCID-5.
6. Able to safely abstain from alcohol for at least 48 hours without requiring medical detox.
7. At Baseline meet DSM-5 criteria for current PTSD with a symptom duration of at least 6 months per the CAPS-5.
8. Are able to swallow pills.
9. Agree to have study visits recorded, including Experimental Sessions, assessments, and non-drug therapy sessions.
10. Able to provide a contact (relative, spouse, close friend, or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming unwell or unreachable.
11. Able to identify an appropriate support person to stay with the participant on the evenings of the Experimental Sessions.

    Weight
12. Body Mass Index (BMI) in the range of 18-35. Sex and Contraceptive/ Barrier Requirements
13. For participants assigned female sex at birth:

    -A participant is eligible to participate if not pregnant, not planning to become pregnant, or is not breastfeeding and one of the following conditions applies: oIs not able to become pregnant OR oIs a person able to be pregnant (PABP) and using a contraceptive method that is highly effective, with a failure rate of <1%. The investigator will evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first does of study intervention.

    -A PABP must have a highly sensitive negative urine pregnancy test at study entry and prior to each Experimental Session, see Schedule of Activities.

    Informed Consent
14. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

    Other Inclusions
15. Agree to inform the investigators within 48 hours of any medical conditions and procedures.
16. May have asymptomatic Hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed.
17. May have a history of or current Diabetes Mellitus (Type 2) if additional screening measures of Hemoglobin A1c levels are less than 7, identifying that the Type 2 diabetes is well controlled, if the condition is judged to be stable on effective management, and with approval by the study clinician.
18. May have hypothyroidism if taking adequate and stable thyroid replacement medication.
19. May have a history of, or current, glaucoma if approval for study participation is received from an ophthalmologist.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Have symptomatic liver disease or have significant liver enzyme elevations.

   1. Alanine transaminase (ALT) or aspartate transaminase (AST) > 3 x upper limit of normal (ULN).
   2. Total bilirubin > 1.5 x ULN or direct bilirubin < 35%.
2. Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.

   a)Note: Stable chronic liver disease (including Gilbert's syndrome, asymptomatic gallstones, and chronic stable hepatitis B (e.g., the presence of hepatitis B surface antigen or positive hepatitis C antibody test result without evidence of active infection at screening or within 3 months prior to starting study intervention) is acceptable if the participant otherwise meets entry criteria.
3. Have a history of seizures or delirium tremens.
4. Significant alcohol withdrawal symptoms, defined as a Clinical Institute Withdrawal Assessment of alcohol scale, revised (CIWA-Ar) >10.
5. Have a recent history of clinically significant hyponatremia or hyperthermia.
6. Have a marked Baseline QTcF interval >450 ms demonstrated on repeated ECG assessments. Participants whose QTcF exceeds this value during screening may be initially enrolled if a pre-study concomitant medication is suspected to be prolonging the QT-interval.

   a)Note: The QTcF is the QT interval corrected for heart rate according to Fridericia's formula. It is either machine-read or manually over-read.
7. Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate. This includes, but is not limited to, a history of myocardial infarction, cerebrovascular accident, heart failure, severe coronary artery disease, or aneurysm.

   a)Participants with other mild, stable chronic medical problems may be enrolled if the study physician and principal investigators agree the condition would not significantly increase the risk of MDMA administration or be likely to produce significant symptoms during the study that could interfere with study participation or be confused with side effects of the study drug.
8. Examples of stable medical conditions that could be allowed include, but are not limited to, Diabetes Mellitus (Type 2), Human Immunodeficiency Virus (HIV) infection, Gastroesophageal Reflux Disease (GERD), hypothyroidism (if taking adequate and stable thyroid replacement medication), glaucoma (if approval for study participation is received from an ophthalmologist).
9. Have a diagnosis of uncontrolled hypertension, defined as repeated blood pressure readings of 140 millimeters of Mercury [mmHg] systolic or 90 mmHg diastolic. The diagnosis may be confirmed by repeated clinic measurements or home blood pressure monitoring if clinically indicated.
10. Have a history of ventricular arrhythmia at any time, other than occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease.
11. Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation.
12. Have a history of arrhythmia, other than premature atrial contractions (PACs) or occasional PVCs in the absence of ischemic heart disease, within 12 months of screening.

    a)Participants with a history of atrial fibrillation, atrial tachycardia, atrial flutter or paroxysmal supraventricular tachycardia or any other arrhythmia associated with a bypass tract may be enrolled only if they have been successfully treated with ablation and have not had recurrent arrhythmia for at least one year off all antiarrhythmic drugs or are under adequate and stable pharmacologic treatment for atrial fibrillation for at least a year, as confirmed by a cardiologist.
13. Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).

    Psychiatric Conditions
14. Have engaged in a new form of psychiatric or mental health care within 12 weeks of enrollment, including Electroconvulsive Therapy (ECT) and ketamine-assisted therapy.
15. Are currently prescribed antidepressant medication (antidepressant pharmacotherapy use considered if assessed by physician and titrated down to 5 half-lives + 1 week washout).
16. Are currently prescribed antipsychotic medications.
17. Are likely, in the investigator's opinion and via observation during the Preparatory Period, to be re-exposed to their index trauma or other significant trauma directly during the study.
18. Have a current moderate (not in early remission in the 3 months prior to enrollment and meets at least 5 of 11 diagnostic criteria per DSM-5) or severe cannabis use disorder within the 12 months prior to enrollment (meets at least 6 of 11 diagnostic criteria per DSM-5).

    a)May have current mild cannabis use disorder (meets 3 of 11 diagnostic criteria per DSM-5) or moderate cannabis use disorder in early remission for the 3 months prior to enrollment (meets 4 or 5 of 11 diagnostic criteria per DSM-5).
19. Have an active substance use disorder (other than cannabis) at any severity within 12 months prior to enrollment.
20. Have used MDMA or Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 12 months of the first Experimental Session
21. Any participant presenting current serious suicide risk, as determined through psychiatric interview, responses to C-SSRS, and clinical judgment of the investigator will be excluded; however, history of suicide attempts is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior, in the judgment of the investigator, will not be enrolled. Any participant presenting with the following on the Baseline C-SSRS will be excluded:

    1. Suicidal ideation score of 4 or greater within the last 6 months of the assessment at a frequency of once a week or more
    2. Suicidal ideation score of 5 within the last 6 months of the assessment
    3. Any suicidal behavior, including suicide attempts or preparatory acts, within the last 6 months of the assessment. Participants with non-suicidal self-injurious behavior may be included if approved by the study physician.
22. Would present a serious risk to others as established through clinical interview and contact with treating providers.

    Prior/Concomitant Therapy
23. Require ongoing concomitant therapy with a psychiatric medication with exceptions described in protocol section on Concomitant Medications (refer to Appendix 3: Permitted and Prohibited Medications).
24. Current use of pharmacotherapies (i.e., naltrexone, acamprosate, or disulfiram) to treat alcohol use.
25. Require use of concomitant medications that could prolong the QT interval during Experimental Sessions.
26. Are currently engaged in trauma-focused psychotherapy or are currently in a treatment program for SUD (self-help programs are not an exclusion).

    Prior/Concurrent Clinical Study Experience
27. Current enrollment in any other clinical study involving an investigational study treatment or any other type of medical research, unless approved by the study team.

    Diagnostic Assessments
28. Have a history of or a current primary psychotic disorder, bipolar affective disorder type I or dissociative identity disorder assessed via the DDIS and clinical interview.
29. Have a current eating disorder with compensatory behaviors.
30. Have current major depressive disorder with psychotic features.
31. Have current Personality Disorders (paranoid, schizoid, schizotypal, antisocial, borderline, histrionic, narcissistic, avoidant, dependent, obsessive-compulsive) assessed via the SCID-5-PD. Diagnoses will be confirmed by clinical interview.

    Other Exclusions
32. Are not able to provide adequate informed consent.
33. Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Principal Investigator or study physician, contraindicates participation in the study.
34. Lack of social support or lack of a stable living situation since the inclusion of a support person to assist the participant following Experimental Sessions is important for ensuring participant safety. If a participant is not able to identify a support person whom the research team may contact, they will not be enrolled.
35. Previous participation in a MAPS/Lykos-sponsored MDMA clinical trial.
36. Employees (and their immediate family members) of MAPS, Lykos, or MAPS Europe B.V; or individuals in a personal relationship with the sponsor investigator.
37. Have any current problem which, in the opinion of the Principal Investigator or study clinician, might interfere with study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2030-05-30 (Estimated)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) total score | from Baseline (Visit 0) to Visit 16 (approximately 22 weeks post-baseline)
  To evaluate the efficacy of MDMA-assisted therapy (MDMA-AT) in reducing PTSD symptom severity in participants with co-occurring PTSD and Alcohol Use Disorder (AUD), as measured by the change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) total score (past 30 days) from Baseline (Visit 0) to Visit 16 (approximately 22 weeks post-baseline). The CAPS-5 total severity score ranges from 0 to 80 with higher scores reflecting worse PTSD symptom severity.

SECONDARY OUTCOMES:
Timeline Follow-Back (TLFB): Drinks per drinking day (past 90 days) | from Baseline (Visit 0) to Visit 16 (approximately 22 weeks post-baseline
  To evaluate the efficacy of MDMA-AT in reducing alcohol use in participants with co-occurring PTSD and Alcohol Use Disorder (AUD), as measured by the change in drinks per drinking day on the Timeline Follow-Back (TLFB; past 90 days) from Baseline (Visit 0) to Visit 16 (approximately 22 weeks post-baseline).
Timeline Follow-Back (TLFB): Number of heavy drinking days (past 90 days) | from Baseline (Visit 0) to Visit 16 (approximately 22 weeks post-baseline
  To evaluate the efficacy of MDMA-AT in reducing alcohol use in participants with co-occurring PTSD and Alcohol Use Disorder (AUD), as measured by the change in the number of heavy drinking days on the Timeline Follow-Back (TLFB; past 90 days) from Baseline (Visit 0) to Visit 16 (approximately 22 weeks post-baseline).
Timeline Follow-Back (TLFB): Percent days abstinent (past 90 days) | from Baseline (Visit 0) to Visit 16 (approximately 22 weeks post-baseline
  To evaluate the efficacy of MDMA-AT in reducing alcohol use in participants with co-occurring PTSD and Alcohol Use Disorder (AUD), as measured by the change in percent days abstinent on the Timeline Follow-Back (TLFB; past 90 days) from Baseline (Visit 0) to Visit 16 (approximately 22 weeks post-baseline).
Inventory of Psychosocial Functioning (IPF) total average score | from Baseline (Visit 0) to Visit 16 (approximately 22 weeks post-baseline
  To assess the impact of MDMA-AT on psychosocial functioning in participants with co-occurring PTSD and Alcohol Use Disorder (AUD), as measured by the change in Inventory of Psychosocial Functioning (IPF) total score (past 30 days) from Baseline (Visit 0) to Visit 16 (approximately 22 weeks post-baseline). Items on the IPF are rated on a 1-7 scale with scales averaged across items; total score range is 1-7. Higher scores reflect worse psychosocial functioning (i.e., greater impariment).

CONTACTS AND LOCATIONS:
Overall Officials: Erica M. Eaton, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Providence VA Medical Center, Providence, RI, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No